CLINICAL TRIAL: NCT05592769
Title: A Pilot Study to Assess the Suitability of the HealthBeacon Injection Care Management System (ICMS) as a Remote Therapeutic Monitoring (RTM) Device for Patients on Injectable Therapy for Respiratory Disease
Brief Title: A Pilot Study to Assess the Suitability of the HealthBeacon Injection Care Management System (ICMS) as a Remote Therapeutic Monitoring (RTM) Device
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: HealthBeacon Plc (Industry)
Collaborators: Modena Allergy & Asthma (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: HBMODENA001
Record Dates: First submitted 2022-10-20; First posted 2022-10-25 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2022-11

CONDITIONS: Respiratory Disease
Keywords: Remote Therapeutic Monitoring; RTM; Severe Asthma; Biologic medication; Injectable medication; Adherence; Compliance; Persistence; Remote monitoring
MeSH Terms: conditions — Respiration Disorders; Asthma; Patient Compliance

STUDY DESIGN:
Intervention Model Description: All participants will be enrolled to the one study arm, in which they will all be provided with access to the HealthBeacon Injection Care Management System (ICMS). Participants will be identified and enrolled from the clinical site by the Study Personnel.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- HealthBeacon Injection Care Management System (ICMS) Arm (Experimental): All participants enrolled will be recruited to this study arm and provided with access to the HealthBeacon ICMS.
  Interventions: Device: HealthBeacon Injection Care Management System (ICMS)

INTERVENTIONS:
Device: HealthBeacon Injection Care Management System (ICMS) — All participants will receive access to the HealthBeacon ICMS to remotely monitor adherence to therapy in the home setting. The system includes the following items/services:
  * The HealthBeacon Smart Sharps Bin
  * The HealthBeacon Companion App
  * HealthBeacon Care Team Support (including smart dose reminders and intervention calls)
  * Waste Management Services
  Participants will also be issued the following interventions to enable collection of the secondary endpoints:
  -Participant Feedback Questionnaire (issued electronically upon study completion, to gather feedback on the HealthBeacon ICMS)

SUMMARY:
This goal of this study is to assess the suitability of the HealthBeacon Injection Care Management System (ICMS) as a Remote Therapeutic Monitoring (RTM) device for patients on injectable medications in the home-setting, for the management of respiratory disorders.

The HealthBeacon ICMS is composed of the Smart Sharps Bin, Companion App and Care Team support. The Smart Sharps Bin a digitally connected sharps container and is pre-programmed with a patient's injection schedule. It creates a time-stamped record of each used injection deposited into it to calculate a patients' adherence to treatment. Following disposal, the next date of injection and rotating injection site is updated without requiring any extra work on behalf of the patient. The system also proactively supports enhanced compliance through a series of smart dose reminders and intervention calls, to help patients stay on track. Clinical teams can then review patient adherence data remotely via an online platform.

The main aims of this study include the following:

* To demonstrate the suitability of the HealthBeacon ICMS as an RTM device for respiratory patients through successful billing and reimbursement for physicians
* To provide data to support the reimbursement of the HealthBeacon ICMS by Private Payors in the future

Participants prescribed injectable medication for the treatment of a diagnosed respiratory condition will be enrolled by the Principal Investigator (PI) and referred to HealthBeacon. Participants will then be provided with access to the HealthBeacon ICMS to remotely track and support their adherence to treatment in the home-setting. Participants will use the system for 6 months and their adherence data during this time will be collected, which the PI and clinical team involved will be able to remotely access and review.

At various stages of the study, the applicable RTM codes will be billed for, for each participant. These stages include when providing each participant with access to the HealthBeacon system, including the Smart Sharps Bin, when providing each participant with education on how to use the device, and when the clinical team monitors each individual patients' adherence data collected by the HealthBeacon system on a monthly basis.

DETAILED DESCRIPTION:
The HealthBeacon ICMS is an adherence support platform for patients on injectable medications in the home-setting. The Smart Sharps Bin electronically records each time a used injection device is deposited into it by means of an infra-red sensor and camera. This data is compared to an individuals' treatment schedule pre-programmed to the unit, to determine the patient's adherence to therapy. The bin also issues reminders to patients when doses are due by means of a blue light on its upper surface. Smart Short Message Service (SMS) dose reminders are also provided to help patients stay on track. The bin displays patients personal adherence score, date of their next injection and at which rotating injection site on a small screen on its upper surface. When a used injection is deposited into the Smart Sharps Bin, patients' adherence automatically updates as does the date of their next injection. This information is also visible for patients to review in the HealthBeacon Companion App (the "App"). Within the App, patients can also tailor their dose reminder preferences, see a log of all doses taken, access educational materials and view their injection schedule details. They may also remotely self-report a dose as taken in the App, if they were away from their Smart Sharps Bin at the time of injection. Patients' adherence data, as collected by the HealthBeacon ICMS, is then available for referring physicians and clinical teams to remotely review, providing teams with greater insight and more accurate information regarding patient compliance. HealthBeacon also remotely monitor the capacity of the Smart Sharps Bins, and provide patients with replacement bins when they reach full capacity whilst arranging collection of full bins through HealthBeacon's mail-back program.

The Centres for Medicare and Medicaid Services (CMS) released the Remote Therapeutic Monitoring (RTM) codes in January 2021 to enable enhanced reimbursement of remote monitoring services. Unlike existing Remote Physiological Monitoring (RPM) codes which required collection of physiological data points, the RTM codes enable reimbursement of devices which monitor therapy adherence, in particular for respiratory and/or musculoskeletal system conditions.

As a remote device to track and support adherence to medications, the HealthBeacon ICMS is well positioned to fulfil the definition of an RTM device. Key steps in the patient referral and usage pathway, including providing access to the HealthBeacon system, initial set up and education on how to use it, and its remote adherence monitoring capabilities, correspond to separate billing events under the RTM codes. Therefore, HealthBeacon believe the system can be successfully implemented as an RTM device with reimbursement for physicians. This study aims to demonstrate this by providing real-world data on patient usage of the system, implementation into clinical practice and primarily by assessing the outcome of the billing process under the RTM codes.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be prescribed an at-home injectable biologic medication for the treatment of a respiratory condition.
* Participants must be able to provide informed consent to participate in the study
* Participants must be Medicare/Medicaid patients
* Participants must be 18 years old or older.
* Participants must have access to a smart phone and be familiar with the use of mobile-phone applications
* Participants must ensure they have a suitable place to store their HealthBeacon Smart Sharps Bin in their home setting, where it can remain plugged into a power source
* Participants must ensure they have network coverage in the area where they will keep their HealthBeacon Smart Sharps Bin

Exclusion Criteria:

* Participants under the age of 18
* Participants who are unable to understand the study, comply with the requirements of the study and provide informed consent to participate in it
* Participants who live somewhere with no/very poor network coverage

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-11-10 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Outcome of billing for the HealthBeacon Injection Care Management System (ICMS) under Remote Therapeutic Monitoring (RTM) reimbursement codes | 1 year
  Data on the outcome of the billing process for the HealthBeacon ICMS as an RTM device for each participant will be collected throughout the study and the rate of successful reimbursement assessed.Data gathered through this process may also include information on the criteria for successful billing and insights into the reimbursement pathway with real-world examples.

SECONDARY OUTCOMES:
Compliance Data | 1 year
  Compliance data to prescribed treatments will be collected, including adherence and persistence data at both an individual and group level.
Participant Feedback | 1 year
  Feedback on the acceptability and utility of the HealthBeacon ICMS will be collected upon completion of each participant's time in the study. Feedback will be collected via electronic questionnaire.
Physician Feedback | 1 year
  Physician feedback on integration of the HealthBeacon ICMS into clinical workflows and benefits of the system as an RTM device for remote monitoring of patient compliance will be collected upon study completion. Feedback will be collected via electronic questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Modena, Dr, Principal Investigator — Principal Investigator
Locations (1):
- Modena Allergy & Asthma, La Jolla, California, United States